CLINICAL TRIAL: NCT01347021
Title: Sacrospinous Colpopexy Versus High Uterosacral Colpopexy in the Treatment of Genital Prolapse Grade III/IV in Women With Uterus
Brief Title: Compare Sacrospinous Fixation Versus High Uterosacral Ligament Fixation for Uterus Vaginal Prolapse III/IV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Responsible Party: sergio brasileiro martins md, unifesp- gynecology session
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: unifespcep0833/05
Record Dates: First submitted 2011-04-25; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2006-05

CONDITIONS: Uterovaginal Prolapse; Prolapse of Vaginal Vault After Hysterectomy; Complete Tear, Sacrospinous Ligament; Uterosacral Ligament; Rupture
Keywords: vaginal colpopexy sacrospinous; vaginal colpopexy uterosacral
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sacrospinous, pelvic prolapse. (Active Comparator): Women with pelvic prolapse grade III/IV were randomly allocated to the sacrospinous colpopexy (25 women) or high uterosacral (26 women)
  Interventions: Procedure: sacrospinous colpopexy versus high uterosacral colpopexy
- uterosacral , pelvic prolapse. (Active Comparator): Women with pelvic prolapse grade III/IV were randomly allocated to the sacrospinous colpopexy (25 women) or high uterosacral (26 women)
  Interventions: Procedure: sacrospinous colpopexy versus high uterosacral colpopexy

INTERVENTIONS:
Procedure: sacrospinous colpopexy versus high uterosacral colpopexy — Women with uterine prolapse grade III or IV were randomly allocated to the sacrospinous colpopexy or high uterosacral colpopexy with vaginal hysterectomy.Before the surgery P-Qol questionnaire were completed and urogynecological examination include de POP-Q system was done. All patients underwent clinical check-ups 1, 6 and 12 months postoperatively. Each check-up included clinical examination and questionnaire.
  Other Names: Sacrospinous ligament fixation(SLF); McCall culdoplasty

SUMMARY:
The purpose of this study is to compare the vaginal sacrospinous colpopexy and high uterosacral colpopexy in the treatment of genital prolapse grade III/IV in women with uterus.

DETAILED DESCRIPTION:
Hysterectomy is often the traditional approach for women with uterovaginal prolapse. However, hysterectomy alone does not address the underlying problem of deficient apical support. Surgical options for patients with apical prolapse include transvaginal suspension procedures using pelvic structures for fixation, such as the sacrospinous ligament or uterosacral ligaments.The objective of this study is to compare the sacrospinous fixation with high uterosacral in the treatment of uterine prolapse POP-Q stage 3 or 4 in terms of recurrence of prolapse,quality of life,complications,post-operative recovery, hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* pelvic prolapse III/IV
* counselling and informed consent

Exclusion Criteria:

* abnormal cervical smears
* abnormal ultrasound findings of uterus or ovaries or abnormal uterine bleeding
* pelvic radiotherapy

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POPQ) at 12 months follow-up | one year
  Quantification of pelvic organ prolapse, according to the Pelvic Organ Prolapse Quantification system (POPQ), as standardized by the International Continence Society.

SECONDARY OUTCOMES:
subjective improvement in quality of life measured by Quality-of-Life Questionnaire (P-QoL)after surgery at 12 months follow-up | one year

CONTACTS AND LOCATIONS:
Overall Officials: Manoel C B Girão, MD, Study Chair — Federal University of São Paulo; Sergio B Martins, md, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Maher C, Feiner B, Baessler K, Glazener CM. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2010 Apr 14;(4):CD004014. doi: 10.1002/14651858.CD004014.pub4. PMID 20393938
- [Derived] Martins SB, Castro RA, Takano CC, Marquini GV, Oliveira LM, Martins Junior PCF, Dias MM, Girao MJBC, Sartori MGF. Efficacy of Sacrospinous Fixation or Uterosacral Ligament Suspension for Pelvic Organ Prolapse in Stages III and IV: Randomized Clinical Trial. Rev Bras Ginecol Obstet. 2023 Oct;45(10):e584-e593. doi: 10.1055/s-0043-1772592. Epub 2023 Nov 9. PMID 37944925
- See also: clik here for more information about this issue - international urogynecology journal — http://iuga.org